CLINICAL TRIAL: NCT05910086
Title: Multimodal Approach to the Intrathecal Catheter for Obstetric Accidental Dural Puncture
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN632022/CHUSTE
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Spinal Anesthetics Causing Adverse Effects in Therapeutic Use
Keywords: Accidental dural puncture; Epidural blood patch; Intrathecal catheter; Postdural puncture headache; Epidural anesthesia; Obstetrics
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients having an accidental dural puncture during the installation of an epidural anesthesia: patients having an accidental dural puncture during the installation of an epidural anesthesia will be included.
  Analysis datas of medical record.
  Interventions: Other: collection of data from the medical record

INTERVENTIONS:
Other: collection of data from the medical record — collection of data from the medical record:
  1. During epidural space puncture = cerebrospinal fluid (CSF) reflux, presence of glucose / strip, saline injection, intrathecal catheter insertion, intrathecal levobupivacaine and sufentanil injection, catheter insertion time, number of punctures, function of the person performing the procedure.
  2. Analgesia and hemodynamics during labor, blood pressure, pulse rate, amount of local anesthetic used, whether emergency cesarean section was performed
  3. Demographic data (age, weight, height, body mass index (BMI))
  4. Post-partum monitoring of decubitus or orthostatic headaches, intensity, any other associated clinical signs
  5. Analgesics used and their efficacy
  6. The use of one or more blood patches, with the volume injected and their efficacy
  7. Identification of the breach during epidural analgesia or after delivery
  8. Call the patient at 1 week to reassess the episode and its consequences.

SUMMARY:
Accidental dural puncture is an uncommon complication of epidural analgesia and can cause postdural puncture headache.

DETAILED DESCRIPTION:
The aim of this study the effectiveness of a protocol implemented in our department, according to the recommendations of good practice, on the reduction of the use of blood patchs in patients who have had an accidental dural puncture during the implementation of their spinal anesthesia, in order to prevent the use of the blood patch. In addition, intensity of headaches is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients having an accidental dural puncture during the installation of an epidural anesthesia

Exclusion Criteria:

* Patients without accidental dural puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having an accidental dural puncture during the installation of an epidural anesthesia will be included.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Number of epidural blood patch | Day: 7
  Collect from medical records.

SECONDARY OUTCOMES:
headache intensity | Day: 7
  Collect from medical records.
Timeframe for blood patching | Day: 0
  Collect from medical records the Timeframe for blood patching
Number of blood patches required | Day: 7
  Collect from medical records.
Safety of the technique by number of adverse event | Day: 7
  Collect from medical record the adverse event (complications).

CONTACTS AND LOCATIONS:
Overall Officials: Pascal MARTIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No